CLINICAL TRIAL: NCT05354895
Title: Study Oxygenating the Brain With Laser Therapy to Increase Mental Functioning in Bipolar Disorder
Brief Title: Oxygenating the Brain With Laser Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Texas at Austin (Other)
Collaborators: Baszucki Brain Research Fund (Other); Milken Institute (Other)
Responsible Party: Principal Investigator, Jorge Almeida, Director, Bipolar Disorder Center | Associate Professor of Psychiatry, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019060106
Record Dates: First submitted 2022-04-14; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention: Transcranial Infrared Laser Stimulation (TILS) (Experimental): Participants receive 10 minutes of TILS treatment to the right prefrontal cortex once a week for 6 weeks. TILS will use an FDA-cleared 1064-nm laser (CG-5000, Cell Gen Therapeutics, LLC, Dallas, TX). The irradiance will be 0.25 W/cm2, and fluence, 60 J/cm2.
  Interventions: Device: Transcranial infrared laser stimulation

INTERVENTIONS:
Device: Transcranial infrared laser stimulation — non-invasive, non-pharmacologic photobiomodulation device

SUMMARY:
Investigating the application of transcranial infrared laser stimulation in individuals with bipolar disorder.

DETAILED DESCRIPTION:
Individuals with bipolar disorder have progressive cognitive decline with repeated mood episodes. This cognitive dysfunction is associated with decreased prefrontal cortex oxygen metabolism, involving cellular respiration in mitochondria. Transcranial infrared laser stimulation (TILS) of the prefrontal cortex uses a near-infrared wavelength of invisible light that penetrates the cortex and improves the ability of mitochondria to use oxygen in the brain. This new technology has been proven safe and is a non-pharmacologic, portable, convenient, and cost-effective form of modulating brain oxygenation using low-level infrared light. This treatment has shown great potential by improving cognitive and mood functioning in controlled human studies by photoactivation of the terminal enzyme in the mitochondrial respiratory chain called cytochrome oxidase (CCO). This mechanism results in unique functional benefits for neurons by stimulating oxygen metabolism. Since bipolar disorder may involve mitochondrial metabolic abnormalities, TILS is a potentially promising intervention. The investigators propose a study among individuals with bipolar disorder in order to 1) elucidate the physiological mechanisms of TILS using non-invasive neuroimaging methods (fNIRS, fMRI and ASL-MRI), and 2) investigate the benefits on people's cognitive functions and symptoms after TILS.

This is open label clinical trial with a single group assignment to treatment for individuals with bipolar disorder. The investigators will investigate if transcranial infrared laser stimulation (TILS) can upregulate brain activity and improve cognition.

ELIGIBILITY:
Inclusion

1. Able to read, speak, and understand English.
2. DSM-5 primary diagnosis of Bipolar Disorder type 1 or 2, by structured clinical interview (SCID-5).
3. Montgomery-Asberg Depression Rating Scale score ≤ 12.
4. Young Mania Rating Scale score ≤ 7.
5. On at least one anti-mania agent at a therapeutic dose for 6 weeks.
6. On stable doses of any standing psychotropics for 6 weeks.
7. Any standing benzodiazepine to a maximum dose equivalent to 22.5 mg oxazepam or 7.5 mg diazepam per day.

Exclusion Criteria:

1. Unable/unwilling to give informed consent.
2. Diagnosed with current primary psychotic disorder (rather than bipolar disorder).
3. Diagnosed with current manic/hypomanic or depressive episode.
4. Moderate to severe substance use disorder within the past 6 months (except nicotine, caffeine, cannabis).
5. Clinically defined major neurological disorder; including, but not limited to, seizure disorder and history of loss of consciousness due to head injury for greater than 10 minutes, or documented evidence of brain injury.
6. Active suicidal intent/plan as detected on screening assessments, or in the investigator's opinion is likely to attempt suicide within the next 6 months.
7. Clinically significant unstable medical condition.
8. If female: pregnant, not using medically acceptable birth control, or currently breastfeeding.
9. Other conditions judged by the investigator that could prevent the participant from completing the study (such as but not limited to, significant physical disability (e.g., hearing/visual deficits) to perform a neutral memory task and/or neuropsychological test battery).

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Perfusion (Pre and Post Intervention) | PRE = ~1 week before first intervention verses POST 1 = Immediately after 1st intervention/ POST 2 = after 6 weeks of TILS treatment
  Compare brain function as measured with arterial spin labelling, functional near infrared spectroscopy pre and post intervention
Changes in Resting State fMRI (Pre and Post Intervention) | PRE = ~1 week before first intervention verses POST 1 = Immediately after 1st intervention/ POST 2 = after 6 weeks of TILS treatment
  Compare brain function as measured with resting state fMRI pre and post intervention
Changes in Resting State functional near-infrared spectroscopy (Pre and Post Intervention) | PRE = ~1 week before first intervention verses POST 1 = Immediately after 1st intervention/ POST 2 = after 6 weeks of TILS treatment
  Compare brain function as measured with near-infrared spectroscopy pre and post intervention
Changes in task-based fMRI (Pre and Post Intervention): cognitive task with emotional distractors | PRE = ~1 week before first intervention verses POST 1 = Immediately after 1st intervention/ POST 2 = after 6 weeks of TILS treatment
  Compare brain function as measured with near-infrared spectroscopy pre and post
Changes in task-based fMRI (Pre and Post Intervention): monetary reward and punishment | RE = ~1 week before first intervention verses POST 1 = Immediately after 1st intervention/ POST 2 = after 6 weeks of TILS treatment
  Compare brain function as measured with near-infrared spectroscopy pre and post

SECONDARY OUTCOMES:
Changes in Composite Score of Cognitive Function | PRE = ~ 1 week before first intervention verses POST after 6 weeks of intervention
  Composite Score of cognitive function measures

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Medical School at the University of Texas, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barrett DW, Davis RE, Siegel-Ramsay JE, Bichlmeier A, Almeida JRC, Gonzalez-Lima F. Cognitive improvement and prefrontal network interactions in individuals with remitted bipolar disorder after transcranial infrared laser stimulation. Front Psychiatry. 2025 Jan 30;16:1547230. doi: 10.3389/fpsyt.2025.1547230. eCollection 2025. PMID 39950176